CLINICAL TRIAL: NCT01728181
Title: A Phase I/II Study of Tivozanib and Erlotinib as Initial Treatment for Metastatic Non-small Cell Lung Cancer Assigned by VeriStrat® Serum Proteomic Evaluation
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Stopped before approval due to ineffective drug
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI59004
Record Dates: First submitted 2012-11-12; First posted 2012-11-16 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Non-small Cell Lung Cancer; Stage IV Disease; EGFR Unknown or Wild-type
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Disease | interventions — tivozanib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase I (Experimental): Will receive Tivozanib and Erlotinib treatment.
  Interventions: Drug: Tivozanib; Drug: Erlotinib
- Phase II Group 1 (Standard of Care) (Other): Group 1: VeriStrat® predicts the chance of no benefit from erlotinib
  • The patient will get standard-of- care
  Interventions: Other: Standard of Care treatment
- Phase II Group 2 (arm 1) (Active Comparator): Group 2: VeriStrat® predicts the chance of benefit from Erlotinib
  • Arm 1: Patient will get the study drugs Erlotinib and Tivozanib
  Interventions: Drug: Tivozanib; Drug: Erlotinib
- Phase II Group 2 (arm 2) (Placebo Comparator): Group 2: VeriStrat® predicts the chance of benefit from Erlotinib
  • Arm 2: Patient will get the study drug erlotinib and placebo
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Tivozanib — The phase I study will test two dose levels of tivozanib (dose level 1: 1.0 mg and dose level 2: 1.5 mg) given daily for 3 consecutive weeks followed by one week break. Based on the phase I results, the dose of tivozanib will be chosen for the phase II study.
  Other Names: AV-951; KRN951
  Arms: Phase I; Phase II Group 2 (arm 1)
Drug: Erlotinib — 150 mg/day for 28 day cycle. No rest period.
  Arms: Phase I; Phase II Group 2 (arm 1); Phase II Group 2 (arm 2)
Other: Standard of Care treatment — This treatment will be determined by the study doctor and is considered standard of care.
  Arms: Phase II Group 1 (Standard of Care)

SUMMARY:
The current trial "A Phase I/II study of Erlotinib +/- Tivozanib as initial treatment for Metastatic Non-small Cell Lung Cancer assigned by VeriStrat® Serum Proteomic Evaluation" will begin by evaluating toxicity for the combination of Tivozanib and Erlotinib to determine a phase II dose. The phase II portion of the study will seek to duplicate the finding of the BEER trial in a selected population of patients with NSCLC with a VeriStrat® Good signature using two oral agents with Tivozanib substituted for bevacizumab. Phase II will be designed as a selection-based randomized trial. Patients with VeriStrat® Good signature will be assigned to EGFR inhibitor therapy with a randomization to Erlotinib plus/minus Tivozanib. Patients with VeriStrat® Poor signature will be assigned to standard of care. Standard-of-care chemotherapy as first treatment at the discretion of patient and physician will be evaluated for response to treatment, survival and repeat VeriStrat® signature.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of non-squamous, non-small cell lung cancer.
* Stage IV disease.
* Age > 18
* If female and of childbearing potential, documentation of negative pregnancy test within 7 days prior to first dose.
* Sexually active women of childbearing potential must agree to use adequate contraceptive measures, while on study and for 30 days after the last dose of study drug. All fertile female subjects (and their partners) must agree to use a highly effective method of contraception. Effective birth control includes (a) intrauterine device (IUD) plus one barrier method; or (b) 2 barrier methods. Effective barrier methods are male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). (Note: Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are not considered effective for this study).
* Able to provide informed consent and have signed an approved consent form that conforms to federal and institutional guidelines.

Additional Phase II Inclusion Criteria:

-No prior treatment for metastatic disease (Phase II ONLY). Patients who received adjuvant systemic chemotherapy are eligible if greater than 6 months has elapsed.

Prior erlotinib treatment is allowed in phase I.

* Performance status of 0-1.
* One disease site meeting RECIST (version 1.1) criteria for measurable or non-measurable disease. Disease sites measured from the CT portion of a combined PET/CT may be used to document measurable disease (Liver or PET findings may be used only for non-measurable disease).

Exclusion Criteria:

* Significant cardiovascular disease, including:

  * Active, clinically symptomatic left ventricular failure.
  * Uncontrolled hypertension: Systolic blood pressure of >140 mmHg or diastolic blood pressure of >90 mmHg on 2 or more antihypertensive medications, documented on 2 consecutive measurements taken at least 24 hours apart.
  * Myocardial infarction, severe angina, or unstable angina within 6 months prior to administration of first dose of study drug.
  * History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation)
  * Cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with anti-arrhythmic medication)
  * Coronary or peripheral artery bypass graft within 6 months of screening.
* Uncontrolled CNS metastases are not allowed; subjects with previously treated brain metastases will be allowed if the brain metastases have been treated, toxicity of radiation has resolved and steroids are no longer required. Leptomeningeal metastases are not allowed.
* Any of the following hematologic abnormalities:

  * Hemoglobin < 9.0 g/dL
  * Absolute neutrophil count (ANC) < 1500 per mm3
  * Platelet count < 100,000 per mm3
  * INR >1.5 or PTT >1.5 × ULN
* Any of the following serum chemistry abnormalities:

  * Total bilirubin > 1.5 × ULN (or > 2.5 × ULN for subjects with Gilbert's syndrome)
  * AST or ALT > 2.5 × ULN (or > 5 × ULN for subjects with liver metastasis)
  * Creatinine > 2.0 × ULN
  * Proteinuria > 3+ by urinalysis or urine dipstick
* Non-healing wound, bone fracture, or skin ulcer.
* Active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis, or other gastrointestinal condition with increased risk of perforation; history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 4 weeks prior to administration of first dose of study drug.
* Serious/active infection or infection requiring parenteral antibiotics.
* Inadequate recovery from any prior surgical procedure or major surgical procedure within 4 weeks prior to administration of first dose of study drug.
* Significant thromboembolic or vascular disorders within 6 months prior to administration of first dose of study drug, including but not limited to:

  * Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
  * Peripheral arterial ischemia > Grade 2 (per CTCAE Version 4.0)
* Significant bleeding disorders within 6 months prior to administration of first dose of study drug, including but not limited to:

  * Hematemesis, hematochezia, melena or other gastrointestinal bleeding > Grade 2 (per CTCAE Version 4.0)
  * Hemoptysis or other pulmonary bleeding (> 1/2 tsp/event over last 3 months not associated with bronchoscopy)
  * Hematuria or other genitourinary bleeding > Grade 2 (per CTCAE Version 4.0)
* Currently active second primary malignancy, including hematologic malignancies (leukemia, lymphoma, multiple myeloma, etc.), other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, and ductal or lobular carcinoma in situ of the breast. Subjects are not considered to have a currently active malignancy if they have completed anti-cancer therapy and have been disease free for >2 years.
* Pregnant or lactating females.
* History of genetic or acquired immune suppression disease such as HIV; subjects on immune suppressive therapy for organ transplant.
* Life-threatening illness or organ system dysfunction compromising safety evaluation.
* Requirement for hemodialysis or peritoneal dialysis.
* Inability to swallow pills, malabsorption syndrome or gastrointestinal disease that severely affects the absorption of tivozanib, major resection of the stomach or small bowel, or gastric bypass procedure.
* Psychiatric disorder or altered mental status precluding informed consent or protocol related testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Safety of combination tivozanib and erlotinib | 36 months
  Phase I- To define the safety (maximum tolerated dose) of Tivozanib when administered in combination with Erlotinib in patients with NSCL cancer.
Overall Survival | 36 months
  Phase II - Overall survival for selection strategy of Erlotinib +/- Tivozanib

SECONDARY OUTCOMES:
Overall Survival for entire population | 36 months